CLINICAL TRIAL: NCT05514340
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase-II Trial to Assess Safety, and Efficacy of Sovateltide in the Treatment of Hypoxic-ischemic Encephalopathy in Neonates
Brief Title: Assess Safety and Efficacy of Sovateltide in Hypoxic-ischemic Encephalopathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmazz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMZ-1620/CT-2.4/2022
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Neonatal Asphyxia; Neonatal Encephalopathy
Keywords: Hypoxic-Ischemic Encephalopathy; Cerebral Asphyxia; Neonatal Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum

STUDY DESIGN:
Intervention Model Description: In sovateltide group, 3 doses of sovateltide, at 0.3 μg/kg body weight will be administered as an intravenous bolus over 1 minute every 3 hours ± 1 hour on day 1, 3, and day 6 (total dose/day: 0.9 µg/kg body weight).
  In control group, 3 doses of equal volume of normal saline will be administered as an IV bolus over 1 minutes every 3 hours ± 1 hour on day 1, 3 and day 6 post randomization.
  In both treatment groups, subjects will be provided the best available standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this double-blind study, the patient and all relevant personnel involved with the conduct and interpretation of the study (including the investigator, investigational site personnel, and the sponsor or designee's staff) will remain blinded to the identity of the Investigational Product (IP) assigned and the randomization codes. The final randomization list will be kept strictly confidential, filed securely by the independent biostatistician, and accessible only to authorized persons as per the sponsor's standard operating procedures until the completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline + Standard of care (Active Comparator): Patients will receive the best available standard of care. Normal saline will be administered as an intravenous bolus over one minute every 3 hours on day 1, day 3, and day 6 post randomizations.
  Interventions: Drug: Normal Saline along with standard treatment
- Sovateltide + Standard of care (Experimental): Patients will receive the best available standard of care. Dose of sovateltide (0.3 µg/kg) will be administered as an intravenous bolus over one minute every 3 hours on day 1, day 3, and day 6 post randomizations.
  Interventions: Drug: Sovateltide along with standard treatment

INTERVENTIONS:
Drug: Normal Saline along with standard treatment — Sovateltide is an endothelin-B receptor agonist. It has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in hypoxic-ischemic encephalopathy patients. In this arm normal saline along with standard treatment will be given for active comparison.
  Other Names: Vehicle
  Arms: Normal Saline + Standard of care
Drug: Sovateltide along with standard treatment — Sovateltide is an endothelin-B receptor agonist. It has the potential to be a first-in-class neuronal progenitor cell therapeutics that is likely to promote quicker recovery and improve neurological outcome in hypoxic-ischemic encephalopathy patients. In this arm sovateltide along with standard treatment will be given for active comparison.
  Other Names: PMZ-1620
  Arms: Sovateltide + Standard of care

SUMMARY:
Sovateltide (PMZ-1620; IRL-1620) is targeted to be used as a "Treatment for hypoxic-ischemic encephalopathy in neonates," which is a life-threatening condition. Sovateltide augments neuronal progenitor cell differentiation and better mitochondrial morphology and biogenesis to activate a regenerative response in the central nervous system. The only treatment for HIE is therapeutic hypothermia with limited success, and studies indicate that sovateltide may be beneficial in these patients.

DETAILED DESCRIPTION:
Neonatal encephalopathy due to perinatal asphyxia is known as hypoxic-ischemic encephalopathy (HIE). HIE is a serious neurological complication affecting premature and full-term neonates, resulting from oxygen deprivation and reduced blood flow to the neonatal brain, leading to neuronal and white matter injury. Currently, no well-established therapies are considered effective for neonatal HIE. The standard of care at present includes supportive management to maintain cerebral perfusion, metabolic balance, and seizure detection and treatment. Currently, the only neuroprotective treatment for HIE is therapeutic hypothermia. However, improvement in patient outcomes following therapy has been moderate, with only 1 in 6 infants benefitting from therapeutic hypothermia.

Additionally, therapeutic hypothermia is time-sensitive, having a narrow therapeutic window wherein therapy must be initiated within 6 hours of delivery to be effective. Timely initiation is also restricted to those neonatal units having adequate equipment and trained staff for therapeutic hypothermia. Death or disability is reported to occur in 55% of infants receiving therapeutic hypothermia. To the best of our knowledge, there is no pharmacotherapy available for the treatment of HIE. Hence, there is a significant unmet medical need.

ETB receptors located widely throughout the CNS are a necessary component of the developing nervous system and also promote neurorestorative processes involving neurogenesis and synaptogenesis. There was an increased expression of neural progenitor markers, NeuroD1 and Double Cortin, and neural markers for mature neurons, NeuN was observed in the sovateltide group compared to vehicle. In addition, Sovateltide increased the expression of presynaptic markers (synapsin1 and synaptophysin) and post-synaptic marker (Postsynaptic Density-95) compared to vehicle. Our results suggest that sovateltide treatment helps recruit and differentiate neural progenitor cells and augments synaptogenesis and endogenous neurorestorative processes.

Sovateltide is a synthetic analog of ET-1 synthesized in 1992 and is a highly specific ETB receptor agonist. We and others have conducted studies to determine the effects of sovateltide upon its interaction with neural ETB receptors and have found that it enhances angiogenesis and neurogenesis and promotes repair and regeneration. This is indicated by neuronal cell proliferation, alleviation of oxidative stress, improvement of neurological and motor functions, and increase in anti-apoptotic markers. In our preclinical study, sovateltide was shown to have neuroprotective effects by promoting repair and regeneration in the brain in a neonatal rat model of HIE. The study showed that sovateltide treatment alone or in combination with hypothermia significantly (p<0.01) increased ETB receptor expression compared to vehicle-treated rat pups. In addition, enhanced VEGF and NGF expression were observed in rat pups treated with Sovateltide alone or in combination with hypothermia compared to vehicle-treated rat pups (p<0.0001, p<0.0001). Sovateltide alone and in combination with hypothermia also demonstrated a significantly reduced number of apoptotic cells compared to the control group. Furthermore, oxidative stress markers, including malondialdehyde, reduced glutathione, and superoxide dismutase was, significantly improved (p<0.0001, p<0.0001, p<0.0001) in those rat pups treated with sovateltide.

Sovateltide was safe and well-tolerated in a Phase I trial (CTRI/2016/11/007509) in healthy human volunteers. In addition, we conducted human studies in patients with cerebral ischemic stroke (NCT04046484, CTRI/2017/11/010654; NCT04047563, CTRI/2019/09/021373), Alzheimer's disease (NCT04052737, CTRI/2017/12/016394), and acute spinal cord injury (NCT04054414, CTRI/2018/12/016667) patients. In summary, about 300 patients have been treated with sovateltide, and no drug-related adverse event has been reported to date.

We plan to conduct a phase II clinical study to evaluate the safety and efficacy of sovateltide therapy along with supportive management in neonates with perinatal asphyxia (HIE). The dose of sovateltide proposed for this phase II study is 0.3µg/kg same as used in the phase II study in ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Either sex with ≥ 36 weeks of gestational age
2. Receiving supportive management for perinatal asphyxia
3. Perinatal depression, based on at least one of the following:

   * Apgar score of <5 at 10 minutes
   * Need for resuscitation (chest compressions or mechanical ventilation) at birth
   * pH <7.00 or base deficit ≥ 16 mmol/liter in the cord or arterial blood within 60 minutes of birth
   * Moderate/severe encephalopathy evident by at least 3 of 6 modified Sarnat criteria, present between 1 to 6 hours of birth.
4. Informed consent by one of the parents or a legal representative

Exclusion Criteria:

1. Gestational age <36 weeks
2. Admitted to hospital 12-hours after birth
3. A genetic or congenital condition that affects neuronal development
4. TORCH infection
5. Neonatal sepsis
6. Complex congenital heart disease
7. Severe dysmorphic feature
8. Microcephaly (head circumference < 2 Standard Deviations below mean for gestational age)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with death or disability (moderate/severe) | 24 months
  Percentage of patients with death or disability (moderate/severe). Severe disability is defined as any of the following: a Bayley composite cognitive score <70, a GMFCS grade of level 3 to 5, hearing impairment requiring hearing aids, or blindness (vision <20/200). Moderate disability is defined as a composite cognitive score 70 - 84, in addition, one or more of the following: GMFCS grade of level 2, unilateral blindness (vision 20/200 in only one eye), or hearing impairment with no amplification/cochlear implant.

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development Scores | 24 months
  Changes in Bayley Scales of Infant and Toddler Development Scores. Cognitive, Language, Motor, Social-Emotional, and General Adaptive Scales Score as assessed by Bayley Scales of Infant and Toddler Development (BSID)TM measured at 6 months after initiation of treatment and then at every 6 months interval.
Disabling cerebral palsy | 24 months
  Change in the proportion of children with disabling cerebral palsy
Seizures | 24 months
  Change in the proportion of patients with seizures. Clinical or electrical seizures at birth, at 6 hours, 12 hours, 24 hours, 48 hours, 72 hours, 7 days, 30 days, 6 months after initiation of treatment, and then at every 6 months interval.
Brain injury | 14 days]
  The number of patients with brain injury (MRI or EEG evidence of brain injury). Abnormal MRI findings based on NICHD neonatal network score within 1 to 2 weeks of initiation of treatment.
Blindness or hearing impairment | 24 months
  Change in the proportion of patients with blindness or hearing impairment
Adverse events | 24 months
  Incidence of sovateltide-related adverse events
Tolerance | 7 days
  The number of patients not receiving complete treatment due to intolerance to sovateltide.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gulati, Study Chair — Chairman and CEO
Locations (4):
- India (4):
  - Father Muller Medical College Hospital, Mangalore, Karnataka
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Niloufer Hospital, Hyderabad, Telangana
  - GSVM Medical College, Kanpur, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No
Results will be communicated and published as manuscript

REFERENCES:
- [Background] Ramos MD, Briyal S, Prazad P, Gulati A. Neuroprotective Effect of Sovateltide (IRL 1620, PMZ 1620) in a Neonatal Rat Model of Hypoxic-Ischemic Encephalopathy. Neuroscience. 2022 Jan 1;480:194-202. doi: 10.1016/j.neuroscience.2021.11.027. Epub 2021 Nov 23. PMID 34826534
- [Background] Ranjan AK, Gulati A. Sovateltide Mediated Endothelin B Receptors Agonism and Curbing Neurological Disorders. Int J Mol Sci. 2022 Mar 15;23(6):3146. doi: 10.3390/ijms23063146. PMID 35328566
- [Background] Gulati A, Agrawal N, Vibha D, Misra UK, Paul B, Jain D, Pandian J, Borgohain R. Safety and Efficacy of Sovateltide (IRL-1620) in a Multicenter Randomized Controlled Clinical Trial in Patients with Acute Cerebral Ischemic Stroke. CNS Drugs. 2021 Jan;35(1):85-104. doi: 10.1007/s40263-020-00783-9. Epub 2021 Jan 11. PMID 33428177
- [Background] Ranjan AK, Briyal S, Gulati A. Sovateltide (IRL-1620) activates neuronal differentiation and prevents mitochondrial dysfunction in adult mammalian brains following stroke. Sci Rep. 2020 Jul 29;10(1):12737. doi: 10.1038/s41598-020-69673-w. PMID 32728189